CLINICAL TRIAL: NCT01863628
Title: Recognition and Early Intervention on Prodrome in Bipolar Disorders: a Longitudinal Prospective Study of the Offspring of Parents With Bipolar Disorder
Brief Title: Recognition and Early Intervention on Prodrome in Bipolar Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Psychiatric Hospital (Other Government)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Guiyun Xu, Associate Professor, Guangzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20120508; 2011B031800154 (Other Grant/Funding Number: Guangdong Science and technology Department)
Record Dates: First submitted 2013-05-21; First posted 2013-05-29 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Bipolar Disorder
Keywords: Prodromal Symptoms; bipolar disorder; Neuropsychological Tests; Magnetic Resonance Imaging; Treatment Outcome; aerobic exercise; psychotherapy
MeSH Terms: conditions — Bipolar Disorder; Prodromal Symptoms | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- psychoeducation (Placebo Comparator): including delivering knowledge on symptoms, discussion of suffering mental difficulties, and general coping techniques
  Interventions: Other: psychoeducation
- aerobic exercise (Experimental): The aerobic exercise would include cycling, jogging, table tennis,and playing badminton for 40 mins at least 3 times per week for 3 months. In each exercise, participants are supposed to exercise to the extent of getting sweaty
  Interventions: Other: aerobic exercise

INTERVENTIONS:
Other: aerobic exercise
  Arms: aerobic exercise
Other: psychoeducation
  Arms: psychoeducation

SUMMARY:
Background and study hypothesis:

Many studies including prospective studies have been demonstrated that a long symptomatic prodromal phase exists prior to the onset of full-brown bipolar disorder, lasting for 9-12 years (Egeland et al., 2000). During the prodromal stage, there are three main clusters of syndromes, including hypomania/mania symptoms, depressive symptoms, and signs of attention deficit hyperactivity disorders (Correll et al., 2007; Tillman et al., 2003; Mantere et al., 2008). Of the hypomania/mania symptoms, decreased sleep, elevated mood, irritability, mood lability, increased energy, and psychomotor agitation are present most frequently. The prodromal depressive symptoms are reported to be depressed mood, anhedonia, insomnia, feelings of worthlessness. Among patients with bipolar disorders, 22.5% reported to comorbid with pediatric ADHD. In addition, some symptoms are considered as non-specific such as decreased functioning, anger outburst, social isolation, and anxiety (Egeland et al., 2000).

Offspring of parents with bipolar disorders are much likely to present prodromal symptoms compared to offspring of healthy parents. In a 10-year longitudinal study using 55 prodromal symptoms checklist, , Egeland et al.(2002) found that 38% offspring of parents with bipolar disorder were considered as at risk compared to 17% in children of healthy parents. In a 15-year follow-up study, Duffy et al.,(2009) found that 32.7% offspring (aged 8-25 years old) of parents with bipolar disorder met the criteria of major mood episode.

Objectives:

One primary objective of this study is to prospectively identify the prodromal stage of bipolar disorder.

Another primary objective is to conduct a randomized, place-controlled trial of aerobic exercise on people who suffering from prodromal symptoms to the extent of significantly impaired function, with attempt at delaying or preventing the onset of a full-blown bipolar disorder.

Design of study and the procedures:

The study will consist of two phases: one-week screening period and a randomized, placebo-controlled, 3-month trial. During the screening period, offspring of parents with bipolar disorder will undergo systematically clinical evaluations. The offspring will be evaluated with clinical symptoms assessing scales, neuropsychological tests, magnetic resonance imaging. During the 3-month trial period, the offspring who meet the inclusion criteria will be randomly assigned to receive treatment of aerobic exercise, placebo, or wait-list group. Psychiatrists are scheduled to assess mood, treatment outcome during the 3-month trial.

Subjects and treatment It is expected that 120 offspring of parents with bipolar disorder aged between 10-25 years, meeting the inclusion of prodromal stage, will be included in the study. All of the offspring will undertake the Kiddie Sads Present and Lifetime Version (K-SADS-PL), and a 70 checklist items of potential prodromal symptoms suggest by us as well as by Dr. Correll et al. (2007). The parents of these offspring are to have a DSM-IV (Diagnostic and Statistical Manual of Mental Disorders)-defined bipolar disorder (bipolar I or II), confirmed by the Chinese version of Structured Clinical interview for DSM-IV-TR Axis I Disorders patient edition (SCID-I/P) [First et al., 2002]. The offspring are to be recruited through the referrals by their parents who will receive psychiatric services in the Guangzhou psychiatric Hospital.

The offspring will be randomly assigned to aerobic exercise and placebo controlled groups. The aerobic exercise would include cycling, jogging,table tennis, and playing badminton for 40 mins at least 3 times a week for 3 months. In each exercise, participants are supposed to exercise to the extent of getting sweaty. In the placebo group, participants will receive general psychoeducation, including delivering knowledge on symptoms, discussion of the suffering mental difficulties, and general coping techniques.

Significance:

Bipolar disorder is a common, chronic, and recurrent mental disorder. The recognition of prodromal stage of bipolar disorder and the early intervention on it may help delay or prevent the onset of bipolar disorder.

DETAILED DESCRIPTION:
Background and study hypothesis:

Bipolar disorder is one of the most common recurrent mental illnesses, with a lifetime prevalence of 3.9%, causing physical as well as mental disabilities. Nearly 40% of people with bipolar disorder experience at least one attempt of suicide, and around 10% end up with suicide completed. The mean age of onset for bipolar disorder is 20 years old, and the peak age of onset is between 15 and 19 years. Evidence shows that the first symptom could present in child as early as 3 years old, however, getting a proper diagnosis and treatment for bipolar disorder is delayed for 16.3 years in those presenting the first psychiatric symptom between 3-15 years, and for 9.9 years in those presenting the first psychiatric symptom between 16-25 years. Such a delay compromises largely the treatment as well as functional outcome of bipolar disorders.

Many studies including prospective studies have been demonstrated that a long symptomatic prodromal phase exists prior to the onset of full-brown bipolar disorder, lasting for 9-12 years. During the prodromal stage, there are three main clusters of syndromes, including hypomania/mania symptoms, depressive symptoms, and signs of attention deficit hyperactivity disorders. Of the hypomania/mania symptoms, decreased sleep, elevated mood, irritability, mood lability, increased energy, and psychomotor agitation are present most frequently. The prodromal depressive symptoms are reported to be depressed mood, anhedonia, insomnia, feelings of worthlessness. Among patients with bipolar disorders, 22.5% reported to comorbid with pediatric ADHD. In addition, some symptoms are considered as non-specific such as decreased functioning, anger outburst, social isolation, and anxiety.

Offspring of parents with bipolar disorders are much likely to present prodromal symptoms compared to offspring of healthy parents. In a 10-year longitudinal study using 55 prodromal symptoms checklist, , Egeland et al., found that 38% offspring of parents with bipolar disorder were considered as at risk compared to 17% in children of healthy parents. In a 15-year follow-up study, Duffy et al., found that 32.7% offspring (aged 8-25 years old) of parents with bipolar disorder met the criteria of major mood episode.

Objectives:

One primary objective of this study is to prospectively identify the prodromal stage of bipolar disorder.

Another primary objective is to conduct a randomized, place-controlled trial of aerobic exercise on people who suffering from prodromal symptoms to the extent of significantly impaired function, with attempt at delaying or preventing the onset of a full-blown bipolar disorder.

Design of study and the procedures:

The study will consist of two phases: one-week screening period and a randomized, placebo-controlled, 3-month trial. During the screening period, offspring of parents with bipolar disorder will undergo systematically clinical evaluations. The offspring will be evaluated with clinical symptoms assessing scales, neuropsychological tests, magnetic resonance imaging. During the 3-month trial period, the offspring who meet the inclusion criteria will be randomly assigned to receive treatment of aerobic exercise, placebo, or wait-list group. Psychiatrists are scheduled to assess mood and treatment outcome during the 3-month trial.

Subjects and treatment:

It is expected that 120 offspring of parents with bipolar disorder aged between 10-25 years, meeting the inclusion of prodromal stage, will be included in the study. All of the offspring will undertake the Kiddie Sads Present and Lifetime Version (K-SADS-PL), and a 70 checklist items of potential prodromal symptoms suggested by us as well as by Dr. Correll and his colleagues. The parents of these offspring are to have a DSM-IV (Diagnostic and Statistical Manual of Mental Disorders)-defined bipolar disorder (bipolar I or II), confirmed by the Chinese version of Structured Clinical interview for DSM-IV-TR Axis I Disorders patient edition (SCID-I/P). The offspring are to be recruited through the referrals by their parents who will receive psychiatric services in the Guangzhou psychiatric Hospital.

The offspring will be randomly assigned to aerobic exercise and placebo controlled group. The aerobic exercise would include cycling, jogging, table tennis,and playing badminton for 40 mins at least 3 times a week for 3 months. In each exercise, participants are supposed to exercise to the extent of getting sweaty. In the placebo group, participants will receive general psychoeducation, including delivering knowledge on symptoms, discussion of suffering mental difficulties, and general coping techniques.

Significance:

Bipolar disorder is a common, chronic, and recurrent mental disorder. The recognition of prodromal stage of bipolar disorder and the early intervention on it may help delay or prevent the onset of bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* have at least one biological parent diagnosed as bipolar disorder (bipolar I or II)
* have at least one of the following syndromes i) two or more DSM-IV defined hypomania/mania symptoms, lasting for at least 4 days; ii) two or more DSM defined major depressive symptoms, lasting for 1 week; iii) at least one of the psychotic symptoms, lasting at least 10 min for each manifestation, and 2-7 manifestations a week for at least 3 months, including: ideas of reference; odd ideas, odd belief, unusual perceptual experiences, bizarre thought or speech, Grandiosity, suspicious ideas, paranoid idea, odd mannerisms, hallucination, disorganized/catatonic behavior; iv)two or more of the DSM-IV defined Attention deficit hyperactivity disorder (ADHD)symptoms; and there must be clear evidence of clinically significant impairment in social, academic, or occupational functioning due to ADHD symptoms

Exclusion Criteria:

* DSM-IV defined Axis I disorders;
* Serious general medical illness;
* mental retardation;
* was/is treated with antipsychotic drugs;
* unable to complete neuropsychological tests due to physical conditions;
* in pregnancy and lactation;
* was taking thyroxine therapy in the last three months or is taking hormone therapy

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Clinical Global Impressions (CGI) Scale at 12 weeks | Baseline and 12 weeks
  Clinical Global Impressions (CGI) Scale is used to assess the patient's global functioning prior to and after initiating a study medication. The CGI provides an overall clinician-determined summary measure, taking into account all available information, including a knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function
Diagnostic status | baseline and 3 months after treatment
  to access whether participants are in the defined prodromal stage of bipolar disorder

SECONDARY OUTCOMES:
Change from Baseline in Hamilton Depression Rating Scale at 12 weeks | baseline and after 12 weeks
  Hamilton Depression Rating Scale is used to assess the depressive symptoms.
Change from baseline in Young Mania Rating Scale at 12 weeks | baseline and 12 weeks
  Young Mania Rating Scale is used to assess hypomania/mania symptoms
Change from baseline in Brief Psychiatric Rating Scale at 12 weeks | baseline and 12 weeks
  Brief Psychiatric Rating Scale is used to assess psychotic symptoms.
Change from baseline in Hamilton Anxiety Rating Scale at 12 weeks | baseline and 12 weeks
  Hamilton Anxiety Rating Scale is used to assess anxious symptoms
Change from baseline in Global Assessment Scale at 12 weeks | baseline and 12 weeks
  Global Assessment Scale is a numeric scale (1 through 100) used by mental health clinicians to rate the general functioning of children

OTHER OUTCOMES:
Neuropsychological performance | baseline and 12 weeks
  Neuropsychological performance is valuated with the MATRICS Consensus Cognitive Battery (MCCB), Test of Nonverbal Intelligence, Third Edition (TONI-3), and STROOP task.
  The MATRICS Consensus Cognitive Battery (MCCB), developed by the National Institute of Mental Health (NIMH) Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) initiative, has been recommended as the standard battery for clinical trials of cognition-enhancing interventions for schizophrenia as well as bipolar disorders.
  TONI-3 is used as language free intelligence measure which also helps in the assessment of aptitude, abstract reasoning and problem solving.
Functional magnetic resonance imaging | baseline and 12 weeks
  Functional magnetic resonance imaging or functional MRI (fMRI) is an magnetic resonance imaging procedure that measures brain activity by detecting associated changes in blood flow.
70 prodromal symptoms checklist for bipolar disorder | baseline
  The instrument consists of 70 items assessing different sorts of symptoms, based on the researchers' clinical experiences and the current literature.
70 prodromal symptoms checklist for bipolar disorder | 12 weeks
  The instrument consists of 70 items assessing different sorts of symptoms, based on the researchers' clinical experiences and the current literature.

CONTACTS AND LOCATIONS:
Overall Officials: Guiyun Xu, M.D, Study Director — Guangzhou Psychiatric Hospital; Kangguang Lin, M.D, Principal Investigator — The University of Hong Kong
Locations (2):
- China (2):
  - Guangzhou Psychiatric Hospital, Guangzhou, Guangdong
  - Guangzhou psychiatric Hospital, Guangzhou, Guangdong

REFERENCES:
- [Background] Berk M, Dodd S, Callaly P, Berk L, Fitzgerald P, de Castella AR, Filia S, Filia K, Tahtalian S, Biffin F, Kelin K, Smith M, Montgomery W, Kulkarni J. History of illness prior to a diagnosis of bipolar disorder or schizoaffective disorder. J Affect Disord. 2007 Nov;103(1-3):181-6. doi: 10.1016/j.jad.2007.01.027. Epub 2007 Feb 26. PMID 17324469
- [Background] Correll CU, Penzner JB, Frederickson AM, Richter JJ, Auther AM, Smith CW, Kane JM, Cornblatt BA. Differentiation in the preonset phases of schizophrenia and mood disorders: evidence in support of a bipolar mania prodrome. Schizophr Bull. 2007 May;33(3):703-14. doi: 10.1093/schbul/sbm028. Epub 2007 May 2. PMID 17478437
- [Background] Duffy A, Alda M, Hajek T, Grof P. Early course of bipolar disorder in high-risk offspring: prospective study. Br J Psychiatry. 2009 Nov;195(5):457-8. doi: 10.1192/bjp.bp.108.062810. PMID 19880938
- [Background] Dutta R, Boydell J, Kennedy N, VAN Os J, Fearon P, Murray RM. Suicide and other causes of mortality in bipolar disorder: a longitudinal study. Psychol Med. 2007 Jun;37(6):839-47. doi: 10.1017/S0033291707000347. Epub 2007 Mar 12. PMID 17349107
- [Background] Druss BG, Hwang I, Petukhova M, Sampson NA, Wang PS, Kessler RC. Impairment in role functioning in mental and chronic medical disorders in the United States: results from the National Comorbidity Survey Replication. Mol Psychiatry. 2009 Jul;14(7):728-37. doi: 10.1038/mp.2008.13. Epub 2008 Feb 19. PMID 18283278
- [Background] Egeland JA, Hostetter AM, Pauls DL, Sussex JN. Prodromal symptoms before onset of manic-depressive disorder suggested by first hospital admission histories. J Am Acad Child Adolesc Psychiatry. 2000 Oct;39(10):1245-52. doi: 10.1097/00004583-200010000-00011. PMID 11026178
- [Background] Egeland JA, Shaw JA, Endicott J, Pauls DL, Allen CR, Hostetter AM, Sussex JN. Prospective study of prodromal features for bipolarity in well Amish children. J Am Acad Child Adolesc Psychiatry. 2003 Jul;42(7):786-96. doi: 10.1097/01.CHI.0000046878.27264.12. PMID 12819438
- [Background] Tillman R, Geller B, Bolhofner K, Craney JL, Williams M, Zimerman B. Ages of onset and rates of syndromal and subsyndromal comorbid DSM-IV diagnoses in a prepubertal and early adolescent bipolar disorder phenotype. J Am Acad Child Adolesc Psychiatry. 2003 Dec;42(12):1486-93. doi: 10.1097/00004583-200312000-00016. PMID 14627884
- [Background] Hauser M, Pfennig A, Ozgurdal S, Heinz A, Bauer M, Juckel G. Early recognition of bipolar disorder. Eur Psychiatry. 2007 Mar;22(2):92-8. doi: 10.1016/j.eurpsy.2006.08.003. Epub 2006 Dec 4. PMID 17142013
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Mantere O, Suominen K, Valtonen HM, Arvilommi P, Isometsa E. Only half of bipolar I and II patients report prodromal symptoms. J Affect Disord. 2008 Dec;111(2-3):366-71. doi: 10.1016/j.jad.2008.03.011. Epub 2008 Apr 28. PMID 18442858
- [Background] First MB, Spitzer RL, Gibbon M, Williams JBW. Structured Clinical Interview for DSM-IV-TR Axis I Disorders-Patient Edition (SCID-I/P, 11/2002 Revision). Biometrics Research Department, New York State Psychiatric Institute, New York.2002.